CLINICAL TRIAL: NCT04773431
Title: Phase I Study to Evaluate Safety of LSCD101(Cultured Autologous Limbal Epithelial Cell Sheet) Transplantation for Limbal Stem Cell Deficiency
Brief Title: Safety Evaluation of LSCD101 Transplantation for Limbal Stem Cell Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CliPS Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSCD101_P1
Record Dates: First submitted 2021-01-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Limbus Corneae; Limbus Corneae Insufficiency Syndrome
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LSCD101 (Cultured Autologous Limbal Epithelial Cell Sheet) transplantation (Experimental): LSCD101 (Cultured Autologous Limbal Epithelial Cell Sheet) is transplanted in the lesion.
  Interventions: Drug: LSCD101 (Cultured Autologous Limbal Epithelial Cell Sheet) transplantation

INTERVENTIONS:
Drug: LSCD101 (Cultured Autologous Limbal Epithelial Cell Sheet) transplantation — LSCD101 (Cultured Autologous Limbal Epithelial Cell Sheet) is transplanted in the lesion.

SUMMARY:
Clinical Study Objective:

To evaluate the tolerability and safety after transplantation of LSCD101 in patients with intractable limbal stem cell deficiency

Study Method:

Subjects who finally meet the inclusion/exclusion criteria results of the subject eligibility evaluation will receive transplantation of the investigational product. Adverse drug reaction will be confirmed during 24 weeks after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 or older
* Diagnosed with intractable limbal stem cell deficiency in single eye, with severity in which corneal neovascularization invades more than two quadrants
* No improvement of indication by known treatment (non-surgical/surgical) method according to investigator's judgment
* BCVA 20/40 or less at screening in the eye with the limbal stem cell deficiency
* Voluntarily agreed to participate in this study and signed a consent form

Exclusion Criteria:

* Inappropriate for harvesting limbal epithelial cells for the production of limbal epithelial cell sheet.
* Difficulty in reconstruction of the corneal epithelium because the eye is not closed due to eyelid function problems in the eye with the limbal stem cell deficiency.
* Severe dry eye with problem with tear secretion in both eyes (value of Schirmer I test without anesthesia < 2 mm/5 min at screening)
* Acute ocular surface inflammation of both corneas at Visit 2
* Malignant tumor history (except in case of no recurrence more than 5 years after surgery)
* Uncontrolled comorbidities such as moderate to severe infections and bleeding
* Positive for virus infection (HBV, HCV, HIV, CMV, HTLVⅠ/Ⅱ, syphilis)
* Uncontrolled diabetes (HbA1c ≥9.0%)
* Uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg despite taking antihypertensives at screening)
* Uncontrolled glaucoma (IOP > 21 mmHg despite taking glaucoma medication)
* Pregnant or lactating women
* Women with childbearing potential, those who do not agree to contraception by medically accepted contraceptive methods during clinical trials
* Participation in another clinical study within 4 weeks
* Subjects judged by the investigator to be inappropriate to participate in the clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse event | From limbal tissue collection until 24 weeks after transplantation
  Adverse event

SECONDARY OUTCOMES:
Rate of normal/abnormal results in clinical laboratory test | Before treatment, 1 week, 2 weeks, 4 weeks, 12 weeks, 24 weeks after transplantation
  Comparisons between pre-/post- transplantation are summarized and presented
Blood pressure(systolic/diastolic) at each visit | Before treatment, 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks, 24 weeks after transplantation
  Comparisons between pre-/post- transplantation are summarized and presented.
Pulse rate at each visit | Before treatment, 1 day, 1 week, 2 weeks, 4 weeks, 12 weeks, 24 weeks after transplantation
  Comparisons between pre-/post- transplantation are summarized and presented.
Rate of normal/abnormal results in Electrocardiogram | Before treatment, 4 weeks, 12 weeks, 24 weeks after transplantation
  Comparisons between pre-/post- transplantation are summarized and presented.
Rate of normal/abnormal results in physical examination at each visit | Before treatment, 4 weeks, 12 weeks, 24 weeks after transplantation
  Comparisons between pre-/post- transplantation are summarized and presented.
Rate of eye infection and inflammation | Before treatment, 1 week, 2 weeks, 4 weeks, 12 weeks, 24 weeks after transplantation
  Eye infection and inflammation test (slit lamp microscopy)
Intraocular pressure test | Before treatment, 4 weeks, 12 weeks, 24 weeks after transplantation
  Intraocular pressure test

CONTACTS AND LOCATIONS:
Overall Officials: SoHyang Chung, MD,Ph.D, Principal Investigator — The Catholic University of Korea
Locations (1):
- CliPS, Seoul, South Korea